CLINICAL TRIAL: NCT03008863
Title: Educating Anesthesia Residents to Improve Perioperative Care for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00069462
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Educational Status

ARMS (2):
- Education Intervention (Experimental): The investigators will use an electronic learning (E-learning) curriculum with an educational video and a user-centered checklist for anesthesia residents. This E-learning curriculum will cover how to care for geriatric patients in the preoperative, intraoperative and postoperative settings, and specific interventions that have been shown to improve postoperative outcomes in older patients.
  The checklist will be user-centered. It will remind providers of what they learned in the video and online curriculum, and how to apply these lessons in real-time while they are caring for older patients.
  Interventions: Other: Education
- Control (No Intervention): Residents randomized to this group will receive the current, standard education provided for all Duke Anesthesiology residents.

INTERVENTIONS:
Other: Education
  Arms: Education Intervention

SUMMARY:
1. The investigators will design, test and implement a education curriculum for anesthesia residents teaching geriatric anesthesiology.
2. The investigators will randomize 42 anesthesia residents so that half receive an innovative, e-learning curriculum while the other half receives the current standard curriculum. We will assess their medical knowledge, and the amount of anesthesia delivered to patients after the curriculum is implemented.
3. The investigators will analyze any changes in clinical practice of residents in the care of elderly patients. Enrollment will be voluntary for all residents. Also, the investigators will not interfere with clinical management of any patients by residents which are done under direct supervision of faculty.

ELIGIBILITY:
Inclusion Criteria:

* Duke Anesthesiology Resident
* Willing to comply with study activities and guidelines

Exclusion Criteria:

* Unable to comply with study activities and guidelines

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
average minimum alveolar concentration (MAC) fraction in patients over age 65 given general anesthesia by residents | 6 months

SECONDARY OUTCOMES:
change in residents' geriatric anesthesia knowledge base to be measured using a pre- and post-test | 6 months
mean bispectral index value in patients over age 65 given monitored sedation by residents | 6 months
frequency of use of medications known to increase delirium risk given to patients over age 65 by residents | 6 months
mean doses of medications known to increase delirium risk given to patients over age 65 by residents | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miles Berger, MD, Phd, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Berger M, Eleswarpu SS, Cooter Wright M, Ray AM, Wingfield SA, Heflin MT, Bengali S, Udani AD. Developing a Real-Time Electroencephalogram-Guided Anesthesia-Management Curriculum for Educating Residents: A Single-Center Randomized Controlled Trial. Anesth Analg. 2022 Jan 1;134(1):159-170. doi: 10.1213/ANE.0000000000005677. PMID 34709008